CLINICAL TRIAL: NCT05092919
Title: The Effect of Sweet Flavoring on the Rewarding and Reinforcing Value of Cigarillo Use Among Young Adults
Acronym: FLAV
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Janet Audrain-McGovern, Professor, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 843944
Record Dates: First submitted 2021-09-30; First posted 2021-10-26 (Actual); Results first posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-04

CONDITIONS: Tobacco Use; Cigar Smoking
MeSH Terms: conditions — Tobacco Use; Cigar Smoking | interventions — Flavoring Agents

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Flavor (Other): Either a sweet-flavored or a non-flavored cigarillo
  Interventions: Other: Flavor

INTERVENTIONS:
Other: Flavor — Sweet flavored vs. non-flavored cigarillos.

SUMMARY:
This within-subjects study aims to evaluate the subjective rewarding value, the relative reinforcing value, and the absolute reinforcing value of sweet flavored cigarillos across three separate laboratory visits among 86 young adults (ages 18-24 years old) who have previously smoked > 10 or more cigarillos in their lifetime.

ELIGIBILITY:
Inclusion Criteria:

1. Able to communicate fluently in English (i.e. speaking, writing, and reading).
2. Male and female young adults who are between 18 and 24 years of age who have used > 10 cigarillos in their lifetime.
3. Not currently undergoing smoking cessation treatment or planning to quit smoking cigarettes within the next 30 days.
4. Plan to live in the area for the duration of the study.
5. Willing to use study-provided cigarillos during three laboratory visits.
6. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the combined consent and HIPAA form.

Exclusion Criteria:

Smoking Behavior

1. Use of less than 10 cigarillos in lifetime
2. Current enrollment or plans to enroll in a tobacco cessation program over the duration of the study.
3. Current use of nicotine replacement therapy or other smoking cessation medication.

Alcohol and Drug

1. History of substance abuse (other than nicotine dependence) in the past 12 months and/or currently receiving medical treatment for substance abuse. Counseling and support groups (e.g. Alcoholics Anonymous and Narcotics Anonymous) will not be considered medical treatment for the purposes of this protocol.
2. Current alcohol consumption that exceeds 25 standard drinks/week.
3. Breath alcohol reading (BrAC) greater than .000 at Laboratory Visit 1.
4. Use of e-cigarettes on >5 days in the past 30 days.

Medical

1. Women, including all individuals assigned as "female" at birth, who are pregnant, breast feeding, or planning a pregnancy over the duration of the study period.
2. Serious or unstable disease within the past year (e.g. cancer, heart disease). Applicable conditions will be evaluated on a case-by-case basis by the Principal Investigator.

Psychiatric

1. Lifetime history of schizophrenia or psychosis
2. Lifetime history of a suicide attempt.
3. Current use of medications used to treat mood, such as depression or anxiety.

   1. Individuals will be excluded if they take psychotropic medications that may impact laboratory assessments of nicotine/flavoring reward and reinforcement.
   2. Participants with a history of depression or anxiety will not be excluded- however, participants who are currently taking any medications used to treat these will be ineligible to participate.
   3. Participants who are not currently taking these medications but are receiving treatment such as therapy or counseling will be eligible to participate.
4. Current or recent use of anti-psychotic medications.

General Exclusion

1. Past, current, anticipated, or pending enrollment in another research program over the study period that could potentially impact subject safety, study data, and/or the study design as determined by the Principal Investigator.
2. Any medical condition, illness, disorder, adverse event (AE), or concomitant medication that could compromise participant safety or significantly impact study performance as determined by the Principal Investigator. Subjects may be deemed ineligible for any of the aforementioned reasons at any point throughout the study, as well as during the initial telephone screen.
3. Significant non-compliance with protocol and/or study design as determined by the Principal Investigator. Subjects may be deemed ineligible at any point throughout the study.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Audrain-McGovern J, Manikandan D, Koita F, Klapec O, Pickworth WB, Stone MD. Effect of sweet flavouring on the rewarding and reinforcing value of cigarillo use among young adults. Tob Control. 2025 May 15;34(3):294-301. doi: 10.1136/tc-2023-058307. PMID 38050181

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Flavor
Started | 95
Completed | 86
Not Completed | 9
Not completed — Lost to Follow-up | 7
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: A total of 95 adults reporting cigarillo use attended the baseline visit and enrolled in the study. Among these, 9 participants were excluded from the analysis; 2 participants withdrew from the study due to lack of interest and time commitment issues, while 7 did not attend all three visits, leaving 86 participants to comprise the analytic sample.
Arm/Group | Flavor
Number analyzed (Participants) | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.23 (1.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 63
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 33
  Black/African American | 29
  Other | 24
Cigarillo Use [Count of Participants; unit: Participants] — Cigarillo use was measured at baseline and included a frequent (use in the past day or week) and infrequent (use in the past month or greater) cigarillo use indicator.
  Participants
    Infrequent | 58
    Frequent | 28
Cigarillo Flavor Preference [Count of Participants; unit: Participants] — Cigarillo flavor preference was ascertained by asking 'During the day(s) that you smoked cigarillos, how often were they flavored?' with response options dichotomized into flavor ('Most of the time/Always') and non-flavored ('Sometimes/Rarely/Never') binary indicator.
  Participants
    Non-flavored | 23
    Flavored | 63
Cigarette Use [Count of Participants; unit: Participants] — Use of combustible cigarettes was ascertained by indicators of frequent (use in the past day or week), infrequent (use in the past month or greater), and never (no lifetime use).
  Participants
    Never | 21
    Infrequent | 43
    Frequent | 22
Blunt Use [Count of Participants; unit: Participants] — A blunt is made by taking out some or all of the tobacco in a cigarillo and replacing it with marijuana. The use of cigarillos for blunts was measured and differentiated from cigarillo tobacco use as intended. Blunt use was ascertained by indicators of frequent (use in the past day or week), infrequent (use in the past month or greater), and never (no lifetime use).
  Participants
    Never | 9
    Infrequent | 41
    Frequent | 36
Flavored Risk Perceptions [Mean (Standard Deviation); unit: units on a scale] — Risk perceptions of flavored cigarillo use were measured with an average sum of two items (i.e., 'Flavored cigarillos are less harmful than non-flavored cigarillos' and 'Flavored cigarillos are less addictive than non-flavored cigarillos.') with Likert-style scaling (0=not at all to 6=extremely). The minimum score is 0 and the maximum is 6. Higher scores indicate lower risk perceptions.
  units on a scale | 1.41 (0.61)
Cigarillo Dependence [Mean (Standard Deviation); unit: units on a scale] — The HONC (hooked on nicotine checklist) adapted for cigarillo use is a 10-question checklist with higher scores indicating greater loss of autonomy and the onset of cigarillo dependence. Responses were scored by tallying the number of yes responses (yes=1 and no=0). Cigarillo dependence can range from 0 (low) to 10 (high).
  units on a scale | 1.71 (2.26)
Advertising Exposure [Mean (Standard Deviation); unit: units on a scale] — Exposure to cigarillo advertising and marketing practices was measured with items adapted from PATH and prior research. A composite cigarillo advertising exposure averaged (α=.71) the 10 items which evaluated the type (flavor and non-flavored), frequency, and source (e.g., Internet, television, newspaper, retail stores, or outdoor locations) of exposure on a 5-point Likert type scale (1=never to 5=always).
  units on a scale | 3.24 (1.21)
Receives Marketing Promotions [Count of Participants; unit: Participants] — Exposure to cigarillo advertising and marketing practices was measured with items adapted from PATH and prior research. Exposure to cigarillo promotions included a binary variable indicating any receipt (yes/no) of any type (mail, email, text, or another way) of cigarillo promotional material (e.g., giveaways, direct mail and e-mail coupons, links to online vendors, branded merchandise, celebrity endorsement, music event sponsorship).
  Participants | 12
E-cigarette Use [Count of Participants; unit: Participants] — Use of e-cigarettes was ascertained by indicators of frequent (use in the past day or week), infrequent (use in the past month or greater), and never (no lifetime use).
  Participants
    Never | 19
    Infrequent | 51
    Frequent | 16

OUTCOME MEASURES:

1. Primary Outcome: Subjective Rewarding Value of Cigarillo Flavoring
Description: Subjective rewarding value of cigarillo flavoring will be measured with the Cigarette Evaluation Scale (CES) adapted for cigarillo use. The CES is an 11 item Likert-format (1=not at all to 7=extremely) self-report instrument with established validity and reliability (α > .80). The investigators will focus on the sum of the two-item satisfaction subscale ("Was it satisfying?" and "Did it taste good?") to calculate the subjective rewarding value. The minimum possible score is 2 and the maximum is 14. Higher scores denote greater subjective rewarding value. Primary Outcome measured at visit 1.
Time Frame: Laboratory visit 1 (Day 1, 1.5 hours)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Flavor
Number analyzed (Participants) | 86
score on a scale
  Citrus "Jazz" | 4.03 (1.47)
  Cream | 3.63 (1.42)
  Non-flavored | 3.30 (1.61)

2. Primary Outcome: Relative Reinforcing Value of Cigarillo Flavoring
Description: Relative reinforcing value of cigarillo flavoring will be measured with a validated choice paradigm, evaluating the preference for sweet flavored (the cigarillo with the highest rewarding value measured in visit 1) relative to non-flavored cigarillos. The reinforcement schedule in the non-flavored cigarillo remained constant at a fixed ratio FR-25, while the reinforcement schedule for the sweet-flavored cigarillo increased with a progressive ratio schedule of PR-25x over 10 trials. RRVF will be defined by the breakpoint (highest trial completed across 10 trials to earn puffs for sweet flavored versus non-flavored cigarillos). Higher breakpoints indicate a greater relative reinforcing value. Primary Outcome measured at visit 2.
Time Frame: Laboratory visit 2 (Day 2, 2 hours)
Measure: Mean (95% Confidence Interval); unit: trials
Arm/Group | Flavor
Number analyzed (Participants) | 86
trials
  Sweet flavored | 6.34 [5.98 to 6.70]
  Non-flavored | 3.66 [3.30 to 4.02]

3. Primary Outcome: Absolute Reinforcing Value of Cigarillo Flavoring
Description: Absolute reinforcing value of cigarillo flavoring is operationalized as the number of sweet flavored versus non-flavored cigarillo puffs consumed during the ad libitum smoking session. A research assistant will videotape, monitor, and count the number of cigarillo puffs taken during the 90-minute period. The primary comparison is the amount of consumption (puffs) of the sweet flavored (determined at visit 1) versus non-flavored cigarillo. A greater number of puffs indicates a higher absolute reinforcing value. Primary Outcome measured at visit 3.
Time Frame: Laboratory visit 3 (Day 3, 2.5 hours)
Measure: Mean (95% Confidence Interval); unit: puffs
Arm/Group | Flavor
Number analyzed (Participants) | 86
puffs
  Sweet flavored | 40.88 [37.74 to 44.03]
  Non-flavored | 23.12 [20.25 to 25.98]

ADVERSE EVENTS:
Time Frame: 3 weeks
Description: Serious Adverse Events were defined as any severe or serious medical event definitely related to study participation.
  Adverse Events were defined as any unanticipated medical event definitely related to study participation.
Arm/Group | Flavor
All-Cause Mortality (participants affected / at risk) | 0/86
Serious Adverse Events (participants affected / at risk) | 0/86
Other Adverse Events (participants affected / at risk) | 1/86
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flavor (N=86)
Participant vomited in smoking lab sink after taking cigarillo puffs during Lab visit 2. (General disorders) | 1 (1) — Took 2 cigarillo puffs, felt nauseous then vomited. Attributed it to no food in >12 hours. Reported feeling better after vomiting. Declined to go home, seek medical care, or discontinue participation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-14): https://cdn.clinicaltrials.gov/large-docs/19/NCT05092919/Prot_SAP_000.pdf
  • Informed Consent Form (2022-09-26): https://cdn.clinicaltrials.gov/large-docs/19/NCT05092919/ICF_001.pdf